CLINICAL TRIAL: NCT04498117
Title: A Multicenter Phase 3, Double-Blind, Placebo-Controlled Study Comparing Chemo-Immunotherapy (Paclitaxel-Carboplatin- Oregovomab) vs Chemotherapy (Paclitaxel-Carboplatin- Placebo) in Patients With Advanced Epithelial Ovarian, Fallopian Tube or Peritoneal Carcinoma
Brief Title: Oregovomab Plus Chemo in Newly Diagnosed Patients With Advanced Epithelial Ovarian Cancer Following Optimal Debulking Surgery
Acronym: FLORA-5
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CanariaBio Inc. (Industry)
Collaborators: Gynecologic Oncology Group (Network); Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QPT-ORE-005; GOG-3035 (Other: Gynecologic Oncology Group); FLORA-5 (Other: CanariaBio Inc.); FLORA5 (Other: CanariaBio Inc.)
Record Dates: First submitted 2020-07-28; First posted 2020-08-04 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Carcinoma, Ovarian Epithelial; Ovarian Neoplasms; Ovarian Cancer; Ovarian Serous Adenocarcinoma; Fallopian Tube Neoplasms; Fallopian Tube Adenocarcinoma; Fallopian Tube Serous Adenocarcinoma; Peritoneal Cancer; Peritoneal Carcinoma; Peritoneal Neoplasms
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms | interventions — oregovomab; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1- Surgery Active (Experimental): Six (6) 21-day cycles of chemotherapy with oregovomab given at four (4) cycles (Cycle 1, Cycle 3, Cycle 5, and Cycle 5 plus 12 weeks).
  Interventions: Biological: Oregovomab; Drug: Paclitaxel; Drug: Carboplatin
- Cohort 1 - Primary Surgery Control (Placebo Comparator): Six (6) 21-day cycles of chemotherapy with placebo comparator given with chemotherapy at four (4) cycles (Cycle 1, Cycle 3, Cycle 5, and Cycle 5 plus 12 weeks).
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Biological: Placebo
- Cohort 2 - NACT + Interval Surgery Active (Experimental): In Cohort 2 - NACT + Interval Surgery, subjects must already have received three (3) cycles of paclitaxel and carboplatin neoadjuvant therapy. Subjects in Cohort 2 - NACT + Interval Surgery will receive three (3) cycles of chemotherapy with oregovomab given at four (4) cycles (Cycle 4, Cycle 6, Cycle 6 plus 6 weeks and Cycle 6 plus 18 weeks).
  Interventions: Biological: Oregovomab; Drug: Paclitaxel; Drug: Carboplatin
- Cohort 2 - NACT + Interval Surgery Control (Placebo Comparator): In Cohort 2 - NACT + Interval Surgery, subjects must already have received three (3) cycles of paclitaxel and carboplatin neoadjuvant therapy. Subjects in Cohort 2 - NACT + Interval Surgery will receive three (3) cycles of chemotherapy with placebo comparator given at four (4) cycles (Cycle 4, Cycle 6, Cycle 6 plus 6 weeks and Cycle 6 plus 18 weeks).
  Interventions: Drug: Paclitaxel; Biological: Placebo; Drug: Carboplatin

INTERVENTIONS:
Biological: Oregovomab — 2 mg, dissolved in 2 mL of 0.9% Sodium Chloride Injection USP, then added to 50 mL of Sodium Chloride Injection USP infused over 20 ± 5 minutes
  Other Names: MAb-B43.13
  Arms: Cohort 1- Surgery Active; Cohort 2 - NACT + Interval Surgery Active
Drug: Paclitaxel — 175 mg/m^2, every 3 weeks
  Other Names: Taxol
Drug: Carboplatin — AUC 6 IV Day 1 x 6 cycles (every 21 days)
  Other Names: Paraplatin
  Arms: Cohort 1 - Primary Surgery Control; Cohort 1- Surgery Active
Biological: Placebo — 2 mg, dissolved in 2 mL of 0.9% Sodium Chloride Injection USP, then added to 50 mL of Sodium Chloride Injection USP infused over 20 ± 5 minutes
  Arms: Cohort 1 - Primary Surgery Control; Cohort 2 - NACT + Interval Surgery Control
Drug: Carboplatin — AUC 5-6 IV Day 1 x 6 cycles (every 21 days)
  Other Names: Paraplatin
  Arms: Cohort 2 - NACT + Interval Surgery Active; Cohort 2 - NACT + Interval Surgery Control

SUMMARY:
Study to compare the safety and efficacy of oregovomab versus placebo, administered in combination with specific cycles of a standard six-cycle chemotherapy regimen (paclitaxel and carboplatin), for the treatment of subjects with newly diagnosed advanced ovarian cancer who have undergone optimal debulking.

DETAILED DESCRIPTION:
Phase 3 double-blind, placebo-controlled, multi-center study to compare the safety and efficacy of four administrations of oregovomab 2 mg IV versus placebo, administered in combination with specific cycles of a standard six-cycle chemotherapy regimen (paclitaxel and carboplatin), for the treatment of subjects with newly diagnosed ovarian cancer who have undergone optimal debulking surgery and are either pending initiation of chemotherapy (Cohort 1 - Primary Surgery) or resumption of another three cycles of chemotherapy, having already completed three cycles of neoadjuvant chemotherapy (Cohort 2 - NACT + Interval Surgery).

For Cohort 1 - Primary Surgery, approximately 372 subjects randomized in a 1:1 ratio (i.e., chemotherapy with oregovomab or chemotherapy with placebo). For Cohort 2 - NACT + Interval Surgery, approximately 230 subjects will be randomized in a 1:1 ratio (i.e., chemotherapy with oregovomab or chemotherapy and placebo).

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years old or older.
2. Newly diagnosed epithelial adenocarcinoma of ovarian, fallopian tube or peritoneal origin FIGO Stage III or IV disease.
3. Histologic epithelial cell types: high grade serous adenocarcinoma, high grade endometrioid adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, or adenocarcinoma not otherwise specified (N.O.S.).
4. Completed debulking surgery (either primary debulking surgery or interval debulking surgery at the discretion of the investigator). Debulking surgery must be optimal, R1 or R0 (defined as R1, macroscopic less than 1 cm in diameter, or R0, microscopic or no evidence of tumor). Assessment of debulking surgery will be determined at the time of the surgical procedure, not by post-surgical imaging.

   1. For Cohort 1, subject will undergo primary debulking surgery. Subject must receive initial dose of paclitaxel 175 mg/m^2 given intravenously and carboplatin AUC 6 IV every 3 weeks for 6 cycles. Carboplatin total dose given as 5 consecutive daily pulse doses, for subjects who experiences significant grade 3 or higher emesis. Subsequent dose modifications will be instituted per protocol. Cycle 1 of chemotherapy ± oregovomab/placebo must be anticipated to occur within 6 weeks after primary debulking surgery
   2. For Cohort 2, subject will undergo interval debulking surgery (IDS). Prior to IDS, subjects must have receive 3 cycles of paclitaxel and carboplatin as neoadjuvant treatment. After IDS, subjects must receive paclitaxel 175 mg/m^2 IV and carboplatin AUC 5-6 IV every 3 weeks, starting cycle 4. Cycle 4 of chemotherapy ± oregovomab/placebo must be anticipated to occur within 6 weeks after IDS.
5. Suitable venous access for the study-required procedures
6. Preoperative serum CA-125 levels ≥ 50 U/mL for Cohort 1, serum CA-125 levels ≥ 50 U/mL prior to first neoadjuvant chemotherapy for Cohort 2.
7. Adequate bone marrow function:

   1. Absolute neutrophil count (ANC) ≥ 1,500/µL
   2. Platelets ≥ 100,000/µL
8. Hemoglobin ≥ 8.0 g/dL (Note: Blood transfusion is permitted up to 48 hours before first dose of study treatment).
9. Adequate liver function:

   1. Bilirubin < 1.5 times upper limit normal (ULN)
   2. Lactate Dehydrogenase (LDH), SGOT/AST and SGPT/ALT < 2.5 times ULN
10. Adequate renal function:

    a. Creatinine ≤ 1.5 times ULN
11. ECOG Performance Status of 0 or 1.
12. For women of childbearing potential, must be willing to avoid pregnancy by using highly effective method of contraception from the first dose of study treatment to 6 months after last dose of study treatment as defined per protocol. Belgium and South Korea only: Use of a highly effective method of contraception from 28 days before first dose.
13. Signed informed consent and authorization permitting release of personal health information.
14. Willingness and ability to complete patient quality of life questionnaires.

Exclusion Criteria:

1. BRCA1 or BRCA2 germline gene mutation test result with:

   1. Pathogenic, ambiguous or inconclusive result available within 28 days prior to starting study treatment (subjects with BRCA1 or BRCA 2 variants of uncertain significance can enroll onto the study as long as there is no intent to administer PARP inhibitors for front-line maintenance therapy), or
   2. Known BRCA1 and BRCA2 somatic mutations, if testing is performed
2. Known Somatic Homologous Recombination Deficiency (HRD) who will receive PARP inhibitor front-line maintenance therapy. Subjects with somatic HRD are eligible as long as there is no intent to administer PARP inhibitor front-line maintenance therapy.
3. Subjects with mucinous adenocarcinoma, carcinosarcoma, tumors with neuroendocrine features and low-grade adenocarcinoma.
4. Female subjects who are lactating and breastfeeding, or have a positive serum pregnancy test within 7 days prior to the first dose of study treatment (C1D1 for Cohort 1 or C4D1 for Cohort 2).
5. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
6. Active autoimmune disease, such as rheumatoid arthritis, systemic lupus erythematosus (SLE), ulcerative colitis, Crohn's Disease, multiple sclerosis (MS), or ankylosing spondylitis requiring active disease modifying treatment.
7. Known allergy to murine proteins or hypersensitivity to any of the excipients of the oregovomab, paclitaxel, or carboplatin.
8. Chronically treated with immunosuppressive drugs such as cyclosporine, adrenocorticotropic hormone (ACTH), etc.
9. Chronic therapeutic corticosteroid use, defined as > 5 days of prednisone or equivalent, with the exception of inhalers or those on a pre-planned steroid taper. (Note: Premedication with corticosteroids per institutional standard of care is allowed.)
10. Recognized acquired, hereditary, or congenital immunodeficiency disease, including cellular immunodeficiencies, hypogammaglobulinemia or dysgammaglobulinemia.
11. Clinically significant active infection(s) at the time of screening.
12. Any of the following conditions (on-study testing is not required unless it is required by a specific participating country):

    1. Known HIV-infected subjects unless on effective anti-retroviral therapy with an undetectable viral load within 6 months, or
    2. Known or suspected hepatitis B if active infection (subjects with chronic hepatitis B infection must have an undetectable HBV viral load on suppressive therapy, if indicated; positive surface antibody alone is not an exclusion), or
    3. Known or suspected hepatitis C infection which has not been treated and cured unless currently on treatment with an undetectable viral load).
13. Uncontrolled or life-threatening diseases compromising safety evaluation.
14. Diagnosed or treated for another malignancy within 5 years before the first dose, or previously diagnosed with another malignancy and have any evidence of residual disease including ductal carcinoma in situ of the breast. Subjects with non-melanoma skin cancer, other carcinoma in situ if have undergone complete resection or cervix carcinoma in situ are not excluded if they have undergone complete resection. Synchronous endometrial and prior diagnosis of endometrial cancer within 5 years is not excluded if all of the following conditions are met: Stage IA, superficial myometrial invasion, without lymphovascular invasion, and not poorly differentiated subtypes including papillary serous, clear cell lesions.
15. Contraindications to the use of pressor agents.
16. Undergone more than one surgical debulking or have not recovered from surgery.
17. Anticipated treatment with any other anti-cancer medications, including bevacizumab, PARP inhibitors, or any investigational agent(s) during the study.
18. History or evidence upon physical examination of CNS disease, seizures not controlled with standard medical therapy, or any brain metastases.
19. Any of the following cardiovascular conditions:

    1. Acute myocardial infarction within 6 months before the first dose of study treatment.
    2. Current history of New York Heart Association (NYHA) Class III or IV heart failure.
    3. Evidence of current uncontrolled cardiovascular conditions including cardiac arrhythmias, angina, pulmonary hypertension, or electrocardiographic clinically significant findings.
20. Unable to read or understand or unable to sign the necessary written consent before starting treatment.
21. May not receive any live, attenuated vaccine administered within 28 days (or 4 weeks) prior to enrollment, during the study, and for at least 90 days after the last dose of study treatment.
22. Subjects who receive Hyperthermic Intraperitoneal Chemotherapy (HIPEC), any other anti-cancer medications, including bevacizumab, PARP inhibitors, or any other investigational agent(s) with 3 cycles of paclitaxel and carboplatin neoadjuvant treatment prior to IDS.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 615 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2026-03-26 (Estimated); Study Completion 2028-08-26 (Estimated)

PRIMARY OUTCOMES:
Investigator Assessed Progression Free Survival | Date of randomization until date of first documented disease progression or date of death from any cause, whichever comes first, at up to approximately 6 years.
  Date of randomization to radiographically-confirmed disease progression according to RECIST v1.1 as determined by the investigator or death

SECONDARY OUTCOMES:
Overall Survival | Date of randomization up until date of death from any cause, up to approximately 11 years
  Date of randomization to the date of death
Safety and Tolerability | Date of randomization up until date of discontinuation of treatment, date of significant physical examination changes, date of significant clinical changes, up to approximately 6 years
  Incidence of adverse events (AEs) leading to discontinuation of treatment, frequency/severity of vital signs measurements, physical examination findings, and changes in clinical laboratory parameters
Change in Quality of Life | Changes from baseline assessment, until date of discontinuation, or up to approximately 6 years
  1. Change from baseline in the global health status/QOL scale score of the Functional Assessment of Cancer Therapy-Ovarian (FACT-O TOI)
  2. Three additional questions from the NFOSI-18 in each treatment group

OTHER OUTCOMES:
Efficacy by times to subsequent therapies and time to next progression | Date of randomization, until date of subsequent therapy or death, or up to approximately 6 years
  1. Tumor response measurement by iRECIST
  2. Time to First Subsequent Therapy (TFST), defined as tie form the date of randomization to first subsequent anti-cancer therapy or death
  3. Time to Second Subsequent Therapy, defined as time from the date of randomization to second anti-cancer therapy start date or death
  4. Progression Free Survival 2, defined from the date of randomization to the first documented progression on next-line therapy or death.
Potential Biomarkers | Date of randomization, until date of discontinuation, or up to approximately 6 years
  1. Human Anti-Mouse Antibody (HAMA)
  2. HAMA interference-free CA-125
  3. Neutrophil + Monocyte to Lymphocyte Ratio (NMLR)
  4. Phenotyping or immune subsets, including myeloid-derived suppressor cells (MDSC)
  5. Functional assessment of CD4+ and CD8+ T-cells with a focus on measuring the number and frequency of INF-y-producing CD8+ T-cells using flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Gupta, MD, FRCPC, Study Director — CanariaBio Inc.
Locations (148):
- United States (81):
  - Honor Health, Phoenix, Arizona
  - The University of Arizona Cancer Center, Tucson, Arizona
  - John Muir Health Clinical Research Center, Concord, California
  - Kaiser Permanente Southern California, Irvine, California
  - Moores UC San Diego Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Epic Care, Pleasant Hill, California
  - Kaiser Permanente Riverside Medical Center, Riverside, California
  - University of California, Davis Comprehensive Cancer Center, Sacramento, California
  - Contra Costa Oncology, Walnut Creek, California
  - John Muir Health Gynecologic Cancer Services, Walnut Creek, California
  - University of Colorado Health, Aurora, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Smilow Cancer Hospital, New Haven, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - AdventHealth Orlando, Orlando, Florida
  - Women's Cancer Florida/Women's Cancer Associates, St. Petersburg, Florida
  - Lewis Cancer & Research Pavilion at St. Joseph's Candler, Savannah, Georgia
  - The Queens Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children/University of Hawaii, Honolulu, Hawaii
  - Parkview Research Center, Fort Wayne, Indiana
  - Women's Cancer Care/Mary Bird Perkins Cancer Center, Covington, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - MetroWest Medical Center, Framingham, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Tufts Medical Center Cancer Center in Stoneham, Stoneham, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Minnesota Oncology Hematology - Mercy Hospital, Coon Rapids, Minnesota
  - Minnesota Oncology Hematology, Edina, Minnesota
  - University of Minnesota Health - Maple Grove Clinic, Maple Grove, Minnesota
  - Minnesota Oncology Hematology, Minneapolis, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - Minnesota Oncology Hematology, Saint Paul, Minnesota
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The Valley Hospital (Valley Health), Paramus, New Jersey
  - Womens Cancer Care Associates, Albany, New York
  - Mount Sinai - PRIME, Lake Success, New York
  - Mount Sinai The Blavatnik Family Chelsea Medical Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Montefiore Medical Center PRIME, The Bronx, New York
  - Duke University, Durham, North Carolina
  - Duke Women's Cancer Care Raleigh, Raleigh, North Carolina
  - SCC at UH Geauga Medical Center, Chardon, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Grandview Medical Center/Kettering Medical Center, Kettering, Ohio
  - Cleveland Clinic Hillcrest Hospital, Mayfield Heights, Ohio
  - UH Minoff Health Center - Seidman, Orange, Ohio
  - SCC at St. John's Medical Center, Westlake, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialist and Research Institution, LLC, Tulsa, Oklahoma
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Northwest Cancer Specialists, P.C.-Portland-Rose Quarter, Portland, Oregon
  - Magee Women's Hospital of UPMC, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center at UPMC Passavant, Pittsburgh, Pennsylvania
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - Sanford Research/USD-Sioux Falls, Sioux Falls, South Dakota
  - Texas Oncology, P.A. - Austin, Austin, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - Texas Oncology, P.A. - Fort Worth, Fort Worth, Texas
  - Memorial Herman Hospital, Houston, Texas
  - Texas Oncology San Antonio Medical Center, San Antonio, Texas
  - University of Virginia Health Systems, Charlottesville, Virginia
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Oncology Associates - Hampton, Norfolk, Virginia
  - VCU Massey Cancer Center, Richmond, Virginia
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - MultiCare Regional Cancer Center - Auburn, Auburn, Washington
  - MultiCare Regional Cancer Center-Gig Harbor Medical Park, Gig Harbor, Washington
  - MultiCare Institute for Research and Innovation, Puyallup, Washington
  - MultiCare Regional Cancer Center - Tacoma, Tacoma, Washington
  - University of Wisconsin, Madison, Wisconsin
- Argentina (6):
  - CEMAIC - Centro Medico Privado, Córdoba, Córdoba Province
  - Clínica Universitaria Privada Reina Fabiola, Córdoba, Córdoba Province
  - Sanatorio de la Mujer, Rosario
  - Sanatorio Parque S.A, Salta
  - CER San Juan Centro Polivalente de Asistencia e Inv. Clinica, San Juan
  - Clinicas Viedma S.A., Viedma
- Belgium (3):
  - ZNA Middelheim, Antwerp
  - Cliniques Universitaires Saint-Luc, Brussels
  - Clinique CHC MontLégia, Liège
- Brazil (6):
  - Centro de Pesquisas Clinica Reichow, Blumenau
  - Oncosite - Centro de Pesquisa Clinica e Oncologia, Guimarães
  - Centro Gaucho Integrado de Oncologia, Hematologia, Ensino e Pesquisa - Hospital Mae de Deus, Porto Alegre
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia, Santo André
  - Clínica São Germano - Oncologia, São Paulo
  - Fundação Doutor Amaral Carvalho, São Paulo
- Canada (5):
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - City of Health Hospital at Laval (Cité de la Santé de Laval), Laval, Quebec
  - CHUM Centre de Recherche (affiliated with University of Montreal), Montreal, Quebec
  - McGill University Health Centre/Glen Site/ Royal Victoria Hospital, Montreal, Quebec
  - CHUS - Hôpital Fleurimont, Sherbrooke, Quebec
- Chile (2):
  - Centro de Investigación Clínica Bradford Hill, Santiago
  - Sociedad de Investigaciones Medicas Limitada, Temuco
- Czechia (5):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Bulovka, Prague
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Fakultni nemocnice v Motole, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
- Hungary (5):
  - Del-pesti Centrumkorhaz - Orszagos Hematologiai es Infektologiai Intezet, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Debreceni Egyetem, Debrecen
  - Bacs-Kiskun Megyei Oktatokorhaz, Kecskemét
  - Zala Megyei Szent Rafael Korhaz, Zalaegerszeg
- India (8):
  - Fortis Hospital Ltd, Bangalore
  - Fortis Hospital Ltd, Bengaluru
  - All India Institute of Medical Services, Delhi
  - Max Super Specialty Hospital, Mohali
  - Sushrut Hospital, Mumbai
  - Fortis Hospital, Noida
  - Deenanath Mangeshkar Hospital, Pune
  - Ruby Hall Clinic, Pune
- Italy (3):
  - Azienda Socio Sanitaria Territoriale di Monza (Presidio San Gerardo), Monza
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
  - Università Campus Bio-Medico di Roma, Rome
- Mexico (5):
  - Clinical Medical Research S.C., Orizaba, Veracruz
  - Investigacion Onco Farmaceutica S. de R.L. de C.V. (OncoTech), La Paz
  - Universidad Autonoma de Nuevo Leon, Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey
  - SMIQ S. de R.L. de C.V., Querétaro
  - Centro Potosino de Investigación Medica S.C., San Luis Potosí City
- South Korea (9):
  - National Cancer Center, Goyang
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Soeul
- Spain (5):
  - Hospital Clinic de Barcelona, Barcelona, Catalonia
  - Hospital Universitari Vall d'Hebron, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - ICO l'Hospitalet-Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Instituto Valenciano de Oncologia IVO, Valencia
- Taiwan (5):
  - Taipei Veterans General Hospital, Taipei County, Taipei
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No